CLINICAL TRIAL: NCT00006401
Title: Inhaled NO for the Prevention of Chronic Lung Disease
Brief Title: Inhaled Nitric Oxide for Preventing Chronic Lung Disease in Premature Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 99-233; U01HL064857 (NIH)
Record Dates: First submitted 2000-10-12; First posted 2000-10-13 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Lung Diseases; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Lung Diseases; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Inhaled Nitric Oxide (iNO) (Experimental): Nitric Oxide study gas will be initiated at 5 ppm using the INOvent delivery system. The delivery system provides for masked delivery of the treatment gas. This dose will be used for a 21-day period or until extubation.
  Interventions: Drug: iNO
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: iNO — Inhaled Nitric Oxide for Preventing Chronic Lung Disease in Premature Infants
  Other Names: Inhaled nitric oxide.
  Arms: Inhaled Nitric Oxide (iNO)
Other: Placebo — Inhaled Nitrogen
  Arms: Placebo

SUMMARY:
To determine whether or not inhaled nitric oxide (iNO) safely decreases the incidence of chronic lung disease (CLD) in premature infants.

DETAILED DESCRIPTION:
BACKGROUND:

Despite advances in medical, nursing, and respiratory care, CLD affects up to 50 percent of premature infants. As a result, nearly 50,000 infants in the United States develop CLD. It is desirable to investigate therapies that decrease the incidence of CLD because it is associated with failure to thrive, developmental delay, increased risk of pulmonary infection, reactive airway disease, pulmonary hypertension, and death.

DESIGN NARRATIVE:

This is a randomized, double-blind, placebo-controlled, multi-center study. Three specific hypotheses will be tested: 1) iNO reduces the incidence of CLD; 2) iNO reduces serum and lung (tracheal aspirate) markers of inflammation; and 3) iNO does not increase the incidence of intraventricular hemorrhage in premature neonates. The primary endpoint is survival without CLD (defined as continued oxygen requirement) at 36 weeks post conceptional age.

A total of 793 premature newborns will be enrolled from 14 centers within 48 hours of birth. They will be randomly assigned to receive either placebo or iNO at 5 ppm until the breathing tube can be safely removed or after 21 days. The iNO will be delivered by an INOvent delivery system in such a way that physicians and nurses will not know which treatment each participant is receiving. Management strategies for aspects of patient care including mechanical ventilation, surfactant administration, fluid administration, and steroid use will be determined by physicians at each center. Serial cranial ultrasounds and methemoglobin levels will be monitored to determine adverse events. The first 200 patients will have serial blood samples and tracheal aspirates obtained for measurements of inflammatory mediators, including interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), endothelin-1, myeloperoxidase, neutrophil counts (tracheal aspirates), and endothelin-1 (blood). Participants will be seen at 12 and 24 months of age to monitor the long-term effects on the cardiopulmonary or neurologic systems. At these visits, a health questionnaire will be administered and Bayley II scales of infant development will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Weighing between 500 to 1250 grams at birth
* Gestational age of less than 34 weeks
* Less than 48 hours old
* Respiratory failure on mechanical ventilation
* Absence of structural heart disease (PDA, ASD less than 1 cm, or VSD less than 2 mm are permitted if known prior to study entry)
* Absence of lethal congenital anomaly

Exclusion Criteria:

* Concurrent participation in another experimental study (observational studies will be allowed with prior approval by the Steering Committee and Data and Safety Monitoring Board)
* Active pulmonary hemorrhage
* Unevaluated pneumothorax
* High frequency jet ventilation
* Expected short duration of ventilation (less than 48 hours from birth)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 793 (Estimated)
Dates: Start 2000-09; Primary Completion 2005-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Participant's survival without CLD | (measured at 36 weeks after birth)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Kinsella, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (14):
- United States (14):
  - St. Joseph's Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Univeristy of Southern California/Good Samaritan Hospital, Los Angeles, California
  - Children's Hospital, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Utah Valley Regional Medical Center, Provo, Utah

REFERENCES:
- [Result] Kinsella JP, Cutter GR, Walsh WF, Gerstmann DR, Bose CL, Hart C, Sekar KC, Auten RL, Bhutani VK, Gerdes JS, George TN, Southgate WM, Carriedo H, Couser RJ, Mammel MC, Hall DC, Pappagallo M, Sardesai S, Strain JD, Baier M, Abman SH. Early inhaled nitric oxide therapy in premature newborns with respiratory failure. N Engl J Med. 2006 Jul 27;355(4):354-64. doi: 10.1056/NEJMoa060442. PMID 16870914
- [Derived] Mourani PM, Kinsella JP, Clermont G, Kong L, Perkins AM, Weissfeld L, Cutter G, Linde-Zwirble WT, Abman SH, Angus DC, Watson RS; Prolonged Outcomes after Nitric Oxide (PrONOx) Investigators. Intensive care unit readmission during childhood after preterm birth with respiratory failure. J Pediatr. 2014 Apr;164(4):749-755.e3. doi: 10.1016/j.jpeds.2013.11.062. Epub 2013 Dec 31. PMID 24388320
- [Derived] Watson RS, Clermont G, Kinsella JP, Kong L, Arendt RE, Cutter G, Linde-Zwirble WT, Abman SH, Angus DC; Prolonged Outcomes After Nitric Oxide Investigators. Clinical and economic effects of iNO in premature newborns with respiratory failure at 1 year. Pediatrics. 2009 Nov;124(5):1333-43. doi: 10.1542/peds.2009-0114. Epub 2009 Oct 19. PMID 19841128